CLINICAL TRIAL: NCT02530359
Title: Pirfenidone Effect on the Recovery of Renal Function in Patients With Septic Acute Kidney Injury
Brief Title: Pirfenidone Effect on the Recovery of Renal Function in Septic Acute Kidney Injury
Acronym: AKI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jonathan Samuel Chavez Iñiguez, Nephrologhist, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCGFAA-DRA-PFD
Record Dates: First submitted 2015-06-17; First posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Acute Kidney Injury; Sepsis
Keywords: septic acute kidney injury; pirfenidone
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Active Comparator): Pirfenidone extended release 600mg per mouth every 12 hours for 7 days.
  Interventions: Drug: Pirfenidone extended release
- Group 2 (Active Comparator): Pirfenidone extended release 600mg per mouth in the morning and placebo by night (each treatment every 12 hrs) for 7 days.
  Interventions: Drug: Pirfenidone extended release; Drug: Placebo equivalent
- Group 3 (Placebo Comparator): Placebo equivalent per mouth every 12 hrs for 7 days.
  Interventions: Drug: Placebo equivalent

INTERVENTIONS:
Drug: Pirfenidone extended release — Pirfenidone extended release 600mg per mouth
  Arms: Group 1; Group 2
Drug: Placebo equivalent — Placebo equivalent per mouth
  Other Names: Placebo
  Arms: Group 2; Group 3

SUMMARY:
Patients with Septic AKI will be randomized in three arms, group PFD 1,200 will receive PDF 600mg every 12 hrs per mouth, group PDF 600 will receive PFD 600mg in the morning and placebo equivalent at night and Group Placebo will receive placebo every 12 hrs, all for 7 days, all receive conventional treatment KDIGO guides. We analyze the recovery of renal function as a primary objective.

DETAILED DESCRIPTION:
Septic acute kidney injury (AKI) is the most common cause of AKI in the world, there is no specific treatment for this pathology; the pathophysiology is related to inflammatory pathway and strategies that modulate this are potentially useful. The Pirfenidone (PDF) is an anti-fibrotic and anti-inflammatory treatment, in animal models has shown a beneficial effect on the recovery of renal function immediately after administrated. The investigators propose a triple blind clinical trial,in which septic AKI patients will be randomized in three arms, all receive conventional treatment KDIGO guides, groupPDF 1,200 will receive PDF 600mg every 12 hrs per mouth, group PDF 600 will receive 600mg in the morning and placebo equivalent at night and Group Placebo will receive placebo every 12 hrs, all for 7 days. The Investigators analyze the recovery of renal function as a primary objective, as a secondary objectives clinical variables associated with renal recovery, biochemical variables, inflammatory, molecular variables and measurement of PDF in blood will be analyzed. Patients will be follow-up for 7 days and 28 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

. sepsis

* AKI by serum creatinine, according to the KDIGO guide 2012 Acute Kidney Injury • acute on Chronic kidney disease (baseline creatinine <2 mg / dL)

Exclusion Criteria:

* Chronic kidney disease stage 3b, 4 or 5 (basal serum creatinine > 2mg/dl) known and / or sharpened.

  * chronic dialysis (peritoneal dialysis or hemodialysis)
  * History of AKI and / or RRT in the last three months
  * Pregnancy AKI by other causes other than sepsis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
renal function recovery | within the first 7 days
  serum creatinine in serum <2mg/dl and urinary output >1,200 ml/day
renal function recovery | within the first 28 days
  serum creatinine in serum <2mg/dl and urinary output >1,200ml/day

SECONDARY OUTCOMES:
Urinary Volume | within the first 7 days
  Urinary Volume in milliliters in 24 hours
need of renal replacement therapy (RRT) | within the first 7 days
  the patient still need renal replacement (RRT) by the judgment of the nephrologist.
mortality | within the first 7 days
  the patient dead
serum creatinine levels | within the first 7 days
  serum creatinine levels in mg/dL
serum urea levels | within the first 7 days
  serum urea levels in mg/dL
pirfenidone levels in serum ug/mL | on day 1 and day 7
  pirfenidone levels in serum ug/mL
IL-1 | on day 1 and day 7
  Interleucin 1 in serum pg/mL
IL-6 | on day 1 and day 7
  Interleucin 6 in serum pg/mL
TNF-α | on day 1 and day 7
  tumor necrosis factor in serum pg/dL
Toll-like receptor 4 | on day 1 and day 7
  Toll-like receptor 4 in serum pg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Juan Armenzadriz, Dr, Study Director — Centro Universitario Ciencias de la Salud

REFERENCES:
- [Background] Hsu CY. Where is the epidemic in kidney disease? J Am Soc Nephrol. 2010 Oct;21(10):1607-11. doi: 10.1681/ASN.2010050546. Epub 2010 Sep 2. No abstract available. PMID 20813868
- [Background] Hsu RK, McCulloch CE, Dudley RA, Lo LJ, Hsu CY. Temporal changes in incidence of dialysis-requiring AKI. J Am Soc Nephrol. 2013 Jan;24(1):37-42. doi: 10.1681/ASN.2012080800. Epub 2012 Dec 6. PMID 23222124
- [Background] James M, Pannu N. Methodological considerations for observational studies of acute kidney injury using existing data sources. J Nephrol. 2009 May-Jun;22(3):295-305. PMID 19557705
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Brivet FG, Kleinknecht DJ, Loirat P, Landais PJ. Acute renal failure in intensive care units--causes, outcome, and prognostic factors of hospital mortality; a prospective, multicenter study. French Study Group on Acute Renal Failure. Crit Care Med. 1996 Feb;24(2):192-8. doi: 10.1097/00003246-199602000-00003. PMID 8605788
- [Background] Mehta RL, Pascual MT, Soroko S, Savage BR, Himmelfarb J, Ikizler TA, Paganini EP, Chertow GM; Program to Improve Care in Acute Renal Disease. Spectrum of acute renal failure in the intensive care unit: the PICARD experience. Kidney Int. 2004 Oct;66(4):1613-21. doi: 10.1111/j.1523-1755.2004.00927.x. PMID 15458458
- [Background] Metcalfe W, Simpson M, Khan IH, Prescott GJ, Simpson K, Smith WC, MacLeod AM; Scottish Renal Registry. Acute renal failure requiring renal replacement therapy: incidence and outcome. QJM. 2002 Sep;95(9):579-83. doi: 10.1093/qjmed/95.9.579. PMID 12205335
- [Background] Grams ME, Rabb H. The distant organ effects of acute kidney injury. Kidney Int. 2012 May;81(10):942-948. doi: 10.1038/ki.2011.241. Epub 2011 Aug 3. PMID 21814177
- [Background] Singbartl K, Kellum JA. AKI in the ICU: definition, epidemiology, risk stratification, and outcomes. Kidney Int. 2012 May;81(9):819-25. doi: 10.1038/ki.2011.339. Epub 2011 Oct 5. PMID 21975865
- [Background] Heyman SN, Evans RG, Rosen S, Rosenberger C. Cellular adaptive changes in AKI: mitigating renal hypoxic injury. Nephrol Dial Transplant. 2012 May;27(5):1721-8. doi: 10.1093/ndt/gfs100. PMID 22547749
- [Background] Heyman SN, Rosenberger C, Rosen S. Experimental ischemia-reperfusion: biases and myths-the proximal vs. distal hypoxic tubular injury debate revisited. Kidney Int. 2010 Jan;77(1):9-16. doi: 10.1038/ki.2009.347. PMID 19759527
- [Background] Kinsey GR, Sharma R, Okusa MD. Regulatory T cells in AKI. J Am Soc Nephrol. 2013 Nov;24(11):1720-6. doi: 10.1681/ASN.2013050502. Epub 2013 Oct 17. PMID 24136922
- [Background] Kaushal GP, Shah SV. Challenges and advances in the treatment of AKI. J Am Soc Nephrol. 2014 May;25(5):877-83. doi: 10.1681/ASN.2013070780. Epub 2014 Jan 30. PMID 24480828
- [Background] Nash K, Hafeez A, Hou S. Hospital-acquired renal insufficiency. Am J Kidney Dis. 2002 May;39(5):930-6. doi: 10.1053/ajkd.2002.32766. PMID 11979336
- [Background] Mehta RL. Management of acute kidney injury: it's the squeaky wheel that gets the oil! Clin J Am Soc Nephrol. 2011 Sep;6(9):2102-4. doi: 10.2215/CJN.07720811. Epub 2011 Aug 18. No abstract available. PMID 21852670
- [Background] Yang F, Zhang L, Wu H, Zou H, Du Y. Clinical analysis of cause, treatment and prognosis in acute kidney injury patients. PLoS One. 2014 Feb 21;9(2):e85214. doi: 10.1371/journal.pone.0085214. eCollection 2014. PMID 24586237
- [Background] Akcay A, Turkmen K, Lee D, Edelstein CL. Update on the diagnosis and management of acute kidney injury. Int J Nephrol Renovasc Dis. 2010;3:129-40. doi: 10.2147/IJNRD.S8641. Epub 2010 Sep 29. PMID 21694939
- [Background] Brady HR, Singer GG. Acute renal failure. Lancet. 1995 Dec 9;346(8989):1533-40. doi: 10.1016/s0140-6736(95)92057-9. No abstract available. PMID 7491052
- [Background] Hilton R. Acute renal failure. BMJ. 2006 Oct 14;333(7572):786-90. doi: 10.1136/bmj.38975.657639.AE. No abstract available. PMID 17038736
- [Background] Waikar SS, Curhan GC, Wald R, McCarthy EP, Chertow GM. Declining mortality in patients with acute renal failure, 1988 to 2002. J Am Soc Nephrol. 2006 Apr;17(4):1143-50. doi: 10.1681/ASN.2005091017. Epub 2006 Feb 22. PMID 16495376
- [Background] Chiao H, Kohda Y, McLeroy P, Craig L, Housini I, Star RA. Alpha-melanocyte-stimulating hormone protects against renal injury after ischemia in mice and rats. J Clin Invest. 1997 Mar 15;99(6):1165-72. doi: 10.1172/JCI119272. PMID 9077523
- [Background] Thompson JD, Kornbrust DJ, Foy JW, Solano EC, Schneider DJ, Feinstein E, Molitoris BA, Erlich S. Toxicological and pharmacokinetic properties of chemically modified siRNAs targeting p53 RNA following intravenous administration. Nucleic Acid Ther. 2012 Aug;22(4):255-64. doi: 10.1089/nat.2012.0371. PMID 22913596
- [Background] Sugimoto H, LeBleu VS, Bosukonda D, Keck P, Taduri G, Bechtel W, Okada H, Carlson W Jr, Bey P, Rusckowski M, Tampe B, Tampe D, Kanasaki K, Zeisberg M, Kalluri R. Activin-like kinase 3 is important for kidney regeneration and reversal of fibrosis. Nat Med. 2012 Feb 5;18(3):396-404. doi: 10.1038/nm.2629. PMID 22306733
- [Background] 24. A study to evaluate the safety and efficacy of AC607 for the treatment of kidney injury in cardiac surgery subjects (ACT-AKI).
- [Background] Briguori C, Visconti G, Focaccio A, Airoldi F, Valgimigli M, Sangiorgi GM, Golia B, Ricciardelli B, Condorelli G; REMEDIAL II Investigators. Renal Insufficiency After Contrast Media Administration Trial II (REMEDIAL II): RenalGuard System in high-risk patients for contrast-induced acute kidney injury. Circulation. 2011 Sep 13;124(11):1260-9. doi: 10.1161/CIRCULATIONAHA.111.030759. Epub 2011 Aug 15. PMID 21844075
- [Background] Pickkers P, Heemskerk S, Schouten J, Laterre PF, Vincent JL, Beishuizen A, Jorens PG, Spapen H, Bulitta M, Peters WH, van der Hoeven JG. Alkaline phosphatase for treatment of sepsis-induced acute kidney injury: a prospective randomized double-blind placebo-controlled trial. Crit Care. 2012 Jan 23;16(1):R14. doi: 10.1186/cc11159. PMID 22269279
- [Background] Tumlin J, Wali R, Williams W, Murray P, Tolwani AJ, Vinnikova AK, Szerlip HM, Ye J, Paganini EP, Dworkin L, Finkel KW, Kraus MA, Humes HD. Efficacy and safety of renal tubule cell therapy for acute renal failure. J Am Soc Nephrol. 2008 May;19(5):1034-40. doi: 10.1681/ASN.2007080895. Epub 2008 Feb 13. PMID 18272842
- [Background] Tumlin JA, Chawla L, Tolwani AJ, Mehta R, Dillon J, Finkel KW, DaSilva JR, Astor BC, Yevzlin AS, Humes HD. The effect of the selective cytopheretic device on acute kidney injury outcomes in the intensive care unit: a multicenter pilot study. Semin Dial. 2013 Sep-Oct;26(5):616-23. doi: 10.1111/sdi.12032. Epub 2012 Oct 29. PMID 23106607
- [Background] Faubel S, Chawla LS, Chertow GM, Goldstein SL, Jaber BL, Liu KD; Acute Kidney Injury Advisory Group of the American Society of Nephrology. Ongoing clinical trials in AKI. Clin J Am Soc Nephrol. 2012 May;7(5):861-73. doi: 10.2215/CJN.12191111. Epub 2012 Mar 22. PMID 22442183
- [Background] Taniyama M, Ohbayashi S, Narita M, Nakazawa R, Hasegawa S, Azuma N, Teraoka S, Ota K, Yamauchi S, Margolin SB. Pharmacokinetics of an antifibrotic agent, pirfenidone, in haemodialysis patients. Eur J Clin Pharmacol. 1997;52(1):77-8. doi: 10.1007/s002280050252. No abstract available. PMID 9143872
- [Background] Sutton TA, Fisher CJ, Molitoris BA. Microvascular endothelial injury and dysfunction during ischemic acute renal failure. Kidney Int. 2002 Nov;62(5):1539-49. doi: 10.1046/j.1523-1755.2002.00631.x. PMID 12371954
- [Background] Okusa MD. The inflammatory cascade in acute ischemic renal failure. Nephron. 2002 Feb;90(2):133-8. doi: 10.1159/000049032. PMID 11818695
- [Background] Kinsey GR, Li L, Okusa MD. Inflammation in acute kidney injury. Nephron Exp Nephrol. 2008;109(4):e102-7. doi: 10.1159/000142934. Epub 2008 Sep 18. PMID 18802372
- [Background] Schrier RW, Wang W, Poole B, Mitra A. Acute renal failure: definitions, diagnosis, pathogenesis, and therapy. J Clin Invest. 2004 Jul;114(1):5-14. doi: 10.1172/JCI22353. PMID 15232604
- [Background] Thadhani R, Pascual M, Bonventre JV. Acute renal failure. N Engl J Med. 1996 May 30;334(22):1448-60. doi: 10.1056/NEJM199605303342207. No abstract available. PMID 8618585
- [Background] Star RA. Treatment of acute renal failure. Kidney Int. 1998 Dec;54(6):1817-31. doi: 10.1046/j.1523-1755.1998.00210.x. PMID 9853246
- [Background] Conger JD. Interventions in clinical acute renal failure: what are the data? Am J Kidney Dis. 1995 Oct;26(4):565-76. doi: 10.1016/0272-6386(95)90590-1. PMID 7573008
- [Background] Ronco C, Bellomo R. Prevention of acute renal failure in the critically ill. Nephron Clin Pract. 2003 Jan;93(1):C13-20. doi: 10.1159/000066646. PMID 12411754
- [Background] Kelly KJ, Molitoris BA. Acute renal failure in the new millennium: time to consider combination therapy. Semin Nephrol. 2000 Jan;20(1):4-19. PMID 10651214
- [Background] Shimizu T, Kuroda T, Hata S, Fukagawa M, Margolin SB, Kurokawa K. Pirfenidone improves renal function and fibrosis in the post-obstructed kidney. Kidney Int. 1998 Jul;54(1):99-109. doi: 10.1046/j.1523-1755.1998.00962.x. PMID 9648068
- [Background] Hewitson TD, Kelynack KJ, Tait MG, Martic M, Jones CL, Margolin SB, Becker GJ. Pirfenidone reduces in vitro rat renal fibroblast activation and mitogenesis. J Nephrol. 2001 Nov-Dec;14(6):453-60. PMID 11783601
- [Background] Shihab FS, Bennett WM, Yi H, Andoh TF. Effect of pirfenidone on apoptosis-regulatory genes in chronic cyclosporine nephrotoxicity. Transplantation. 2005 Feb 27;79(4):419-26. doi: 10.1097/01.tp.0000151721.99418.48. PMID 15729167
- [Background] Takakuta K, Fujimori A, Chikanishi T, Tanokura A, Iwatsuki Y, Yamamoto M, Nakajima H, Okada M, Itoh H. Renoprotective properties of pirfenidone in subtotally nephrectomized rats. Eur J Pharmacol. 2010 Mar 10;629(1-3):118-24. doi: 10.1016/j.ejphar.2009.12.011. Epub 2009 Dec 13. PMID 20006961
- [Background] Takakura K, Tahara A, Sanagi M, Itoh H, Tomura Y. Antifibrotic effects of pirfenidone in rat proximal tubular epithelial cells. Ren Fail. 2012;34(10):1309-16. doi: 10.3109/0886022X.2012.718955. Epub 2012 Sep 24. PMID 23002925
- [Background] Chen JF, Ni HF, Pan MM, Liu H, Xu M, Zhang MH, Liu BC. Pirfenidone inhibits macrophage infiltration in 5/6 nephrectomized rats. Am J Physiol Renal Physiol. 2013 Mar 15;304(6):F676-85. doi: 10.1152/ajprenal.00507.2012. Epub 2012 Nov 14. PMID 23152296
- [Background] 46. Hartung J: A note on combining dependent tests of significance. Biometrical J 1999, 41:849-855.
- [Background] Macias-Barragan J, Sandoval-Rodriguez A, Navarro-Partida J, Armendariz-Borunda J. The multifaceted role of pirfenidone and its novel targets. Fibrogenesis Tissue Repair. 2010 Sep 1;3:16. doi: 10.1186/1755-1536-3-16. PMID 20809935
- [Background] Shi S, Wu J, Chen H, Chen H, Wu J, Zeng F. Single- and multiple-dose pharmacokinetics of pirfenidone, an antifibrotic agent, in healthy Chinese volunteers. J Clin Pharmacol. 2007 Oct;47(10):1268-76. doi: 10.1177/0091270007304104. PMID 17906160
- [Background] Cho ME, Kopp JB. Pirfenidone: an anti-fibrotic therapy for progressive kidney disease. Expert Opin Investig Drugs. 2010 Feb;19(2):275-83. doi: 10.1517/13543780903501539. PMID 20050822
- [Background] Panacek EA, Marshall JC, Albertson TE, Johnson DH, Johnson S, MacArthur RD, Miller M, Barchuk WT, Fischkoff S, Kaul M, Teoh L, Van Meter L, Daum L, Lemeshow S, Hicklin G, Doig C; Monoclonal Anti-TNF: a Randomized Controlled Sepsis Study Investigators. Efficacy and safety of the monoclonal anti-tumor necrosis factor antibody F(ab')2 fragment afelimomab in patients with severe sepsis and elevated interleukin-6 levels. Crit Care Med. 2004 Nov;32(11):2173-82. doi: 10.1097/01.ccm.0000145229.59014.6c. PMID 15640628
- [Background] Poltorak A, He X, Smirnova I, Liu MY, Van Huffel C, Du X, Birdwell D, Alejos E, Silva M, Galanos C, Freudenberg M, Ricciardi-Castagnoli P, Layton B, Beutler B. Defective LPS signaling in C3H/HeJ and C57BL/10ScCr mice: mutations in Tlr4 gene. Science. 1998 Dec 11;282(5396):2085-8. doi: 10.1126/science.282.5396.2085. PMID 9851930
- [Background] Chow JC, Young DW, Golenbock DT, Christ WJ, Gusovsky F. Toll-like receptor-4 mediates lipopolysaccharide-induced signal transduction. J Biol Chem. 1999 Apr 16;274(16):10689-92. doi: 10.1074/jbc.274.16.10689. PMID 10196138
- [Background] Samuelsson P, Hang L, Wullt B, Irjala H, Svanborg C. Toll-like receptor 4 expression and cytokine responses in the human urinary tract mucosa. Infect Immun. 2004 Jun;72(6):3179-86. doi: 10.1128/IAI.72.6.3179-3186.2004. PMID 15155619
- [Background] El-Achkar TM, Huang X, Plotkin Z, Sandoval RM, Rhodes GJ, Dagher PC. Sepsis induces changes in the expression and distribution of Toll-like receptor 4 in the rat kidney. Am J Physiol Renal Physiol. 2006 May;290(5):F1034-43. doi: 10.1152/ajprenal.00414.2005. Epub 2005 Dec 6. PMID 16332927
- [Background] Cunningham PN, Wang Y, Guo R, He G, Quigg RJ. Role of Toll-like receptor 4 in endotoxin-induced acute renal failure. J Immunol. 2004 Feb 15;172(4):2629-35. doi: 10.4049/jimmunol.172.4.2629. PMID 14764737
- [Background] Patole PS, Schubert S, Hildinger K, Khandoga S, Khandoga A, Segerer S, Henger A, Kretzler M, Werner M, Krombach F, Schlondorff D, Anders HJ. Toll-like receptor-4: renal cells and bone marrow cells signal for neutrophil recruitment during pyelonephritis. Kidney Int. 2005 Dec;68(6):2582-7. doi: 10.1111/j.1523-1755.2005.00729.x. PMID 16316333
- [Background] Morrell ED, Kellum JA, Hallows KR, Pastor-Soler NM. Epithelial transport during septic acute kidney injury. Nephrol Dial Transplant. 2014 Jul;29(7):1312-9. doi: 10.1093/ndt/gft503. Epub 2013 Dec 29. PMID 24378526
- [Background] Leelahavanichkul A, Yasuda H, Doi K, Hu X, Zhou H, Yuen PS, Star RA. Methyl-2-acetamidoacrylate, an ethyl pyruvate analog, decreases sepsis-induced acute kidney injury in mice. Am J Physiol Renal Physiol. 2008 Dec;295(6):F1825-35. doi: 10.1152/ajprenal.90442.2008. Epub 2008 Oct 15. PMID 18922884
- [Background] Miyaji T, Hu X, Yuen PS, Muramatsu Y, Iyer S, Hewitt SM, Star RA. Ethyl pyruvate decreases sepsis-induced acute renal failure and multiple organ damage in aged mice. Kidney Int. 2003 Nov;64(5):1620-31. doi: 10.1046/j.1523-1755.2003.00268.x. PMID 14531793
- [Background] Chatterjee PK, Yeboah MM, Dowling O, Xue X, Powell SR, Al-Abed Y, Metz CN. Nicotinic acetylcholine receptor agonists attenuate septic acute kidney injury in mice by suppressing inflammation and proteasome activity. PLoS One. 2012;7(5):e35361. doi: 10.1371/journal.pone.0035361. Epub 2012 May 7. PMID 22586448
- [Background] Morrell ED, Kellum JA, Pastor-Soler NM, Hallows KR. Septic acute kidney injury: molecular mechanisms and the importance of stratification and targeting therapy. Crit Care. 2014 Sep 2;18(5):501. doi: 10.1186/s13054-014-0501-5. PMID 25575158
- [Background] Hoste EA, Schurgers M. Epidemiology of acute kidney injury: how big is the problem? Crit Care Med. 2008 Apr;36(4 Suppl):S146-51. doi: 10.1097/CCM.0b013e318168c590. PMID 18382186
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Bagshaw SM, Lapinsky S, Dial S, Arabi Y, Dodek P, Wood G, Ellis P, Guzman J, Marshall J, Parrillo JE, Skrobik Y, Kumar A; Cooperative Antimicrobial Therapy of Septic Shock (CATSS) Database Research Group. Acute kidney injury in septic shock: clinical outcomes and impact of duration of hypotension prior to initiation of antimicrobial therapy. Intensive Care Med. 2009 May;35(5):871-81. doi: 10.1007/s00134-008-1367-2. Epub 2008 Dec 9. PMID 19066848
- [Background] Plataki M, Kashani K, Cabello-Garza J, Maldonado F, Kashyap R, Kor DJ, Gajic O, Cartin-Ceba R. Predictors of acute kidney injury in septic shock patients: an observational cohort study. Clin J Am Soc Nephrol. 2011 Jul;6(7):1744-51. doi: 10.2215/CJN.05480610. PMID 21734090
- [Derived] Chavez-Iniguez JS, Poo JL, Ibarra-Estrada M, Garcia-Benavides L, Navarro-Blackaller G, Cervantes-Sanchez C, Nungaray-Pacheco E, Medina-Gonzalez R, Armendariz-Borunda J, Garcia-Garcia G. Effect of Prolonged-Release Pirfenidone on Renal Function in Septic Acute Kidney Injury Patients: A Double-Blind Placebo-Controlled Clinical Trial. Int J Nephrol. 2021 Jan 13;2021:8833278. doi: 10.1155/2021/8833278. eCollection 2021. PMID 33520317